CLINICAL TRIAL: NCT04770415
Title: Ophthalmic Manifestations of Patients With Mucopolysaccharidosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shrouk Shaban Bakr (Other)
Responsible Party: Sponsor-Investigator, Shrouk Shaban Bakr, Resident doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: mucopolysaccharidosis
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Ophthalmic Manifestations

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mucopolysaccharidosis (MPSs) are a group of disorders caused by inherited defects in lysosomal enzymes resulting in widespread intra- and extra-cellular accumulation of glycosaminoglycan(1,2). They have been subdivided according to enzyme defect and systemic manifestations and include MPS IH (Hurler)(3) , MPS IS (Scheie), MPS IH/S (Hurler/Sheie), MPS II(4,5) (Hunter), MPS III (Sanfilippo)(6) , MPS IV (Morquio)(7,8), MPS VI (Maroteaux-Lamy)(9), MPS VII (Sly)(10,11) and MPS IX (Natowicz)(12). Mucopolysaccharidosis have a spectrum of systemic manifestations, including airway and respiratory compromise, skeletal deformities, intellectual and neurological impairment, cardiac abnormalities, gastrointestinal problems and ocular manifestations(13). Ocular manifestation are common in the mucopolysaccharidosis and may result in significant visual impairment(14). Corneal opacification of varying severity is frequently seen, as well as retinopathy, optic nerve swelling and atrophy, ocular hypertension, and glaucoma(14). New treatment modalities for the systemic manifestations of the mucopolysaccharidosis include bone marrow transplant and enzyme replacement therapy have resulted in an improved prognosis in many cases(15).

ELIGIBILITY:
Inclusion Criteria:

* All patients at any age up to 18 years with any type of MPS confirmed by the enzymatic assay

Exclusion Criteria:

* Any patient other than MPS

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients at any age up to 18 years with any type of MPS
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
early detection and management of ophthalmic manifestations in patients with MPS | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided